CLINICAL TRIAL: NCT06398119
Title: Effect of Visuomotor Training Using Pablo System on Hand Function in Children With Hemiplegic Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Effect of Visuomotor Training Using Pablo System on Hand Function in Children With Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Collaborators: University of Hail (Other)
Responsible Party: Principal Investigator, Shamekh Mohamed El-Shamy, Professor, University of Hail
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Hail University
Record Dates: First submitted 2024-04-28; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Treatment Arm (Active Comparator): The traditional therapy program consisted of one hour provided three times a week for three months. The components of traditional therapy included weight-bearing exercises for the upper limbs, protective extensor push to activate the upper limbs' protective reactions, and passive stretching for the flexors of the wrist and elbow. In order to strengthen the muscles that oppose the spastic muscles, such as the elbow and wrist extensors, various toys were used, along with incentives to motivate the children to complete the exercises. Basic reach, grab, carry, and release techniques, in-hand manipulation techniques, and bilateral hand use are exercises that help with hand abilities.
  Interventions: Other: Traditional Treatment Program; Other: Virtual Reality Program
- Virtual Reality Treatment Arm (Experimental): For virtual reality training, the Pablo system was utilized. In both one- and two-dimensional modules, it is a game-based kind of rehabilitation. Based on the concepts of motor learning, this apparatus is used to train users. Using sensors to operate the games, the Pablo system features several boards, multiball, and handheld devices. The virtual reality program consisted of 45 minutes provided three times a week for three months.
  Interventions: Other: Traditional Treatment Program; Other: Virtual Reality Program

INTERVENTIONS:
Other: Traditional Treatment Program — Traditional Treatment Program for improving hand function
Other: Virtual Reality Program — Virtual Reality Program for improving hand function

SUMMARY:
The aim of this study was to investigate the efficacy of Virtual reality on hand function in Saudi children with hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effect of Virtual reality on hand function in children with hemiplegic CP. Forty children with hemiplegic CP were assigned randomly into two groups (A & B). Control group (A) was received conventional rehabilitation program for the hand. Study group (B) was received conventional rehabilitation program as in group (A) in addition to virtual reality by using the Pablo system.Patients' evaluation was carried out before and after training to assess hand function.

.

ELIGIBILITY:
Inclusion Criteria:

* They had a diagnosis of spastic hemiplegia derived from medical records.
* Scored I-III on the Manual Ability Classification System.
* Not have musculoskeletal disorders that would make it difficult for them to use the VR.
* They had normal or corrected hearing and vision.
* They had no prior experience with the VR.
* They comprehend and follow straightforward instructions to complete the tasks.

Exclusion Criteria:

* They have had upper limb surgery within the last six months.
* They have uncontrollably occurred seizures.
* They have medical conditions that can make using virtual reality dangerous.
* They have attention deficit issues.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline spasticity degrees at 3 months | Baseline and 3 months post-intervention
  Using the Modified Ashworth Scale, the degree of upper limb spasticity was assessed. Based on the degree of muscle resistance felt by the therapist in response to a passive stretch of a joint, this sixfold scale goes from 0 (no spasticity) to 4 (fixed muscle contracture). In this study, the wrist flexor, elbow flexor, and shoulder adductor were examined. In order for the therapist to provide a score, the passive movement was done three times.
Change from baseline grip and pinch strength at 3 months | Baseline and 3 months post-intervention
  Using dynamometry, the strength of the pinch grasp and power were measured and reported in kilograms. A hydraulic hand dynamometer was used to test the power grip strength.The average of the three trials that each participant completed was used for analysis. Every child was instructed to sit on a chair that could be raised or lowered, with a backrest for support, and to keep their head in the middle. They also instructed to flex their hips and knees to a 90-degree angle and keep their feet flat on the ground. With the forearm halfway between supination and pronation, the elbow joint flexed 90 degrees, and the wrist joint in a neutral posture, the arm was positioned next to the torso. Next, the participant was instructed to grasp the dynamometer handle and squeeze it as hard as possible before letting go of it.

CONTACTS AND LOCATIONS:
Overall Officials: Shamekh M Elshamy, Ph.D., Principal Investigator — Professor
Locations (1):
- Maternity and Children Hospital, Ha'il, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No